CLINICAL TRIAL: NCT00202319
Title: Evaluating the Effectiveness of Protocol Directed Sedation Management With Non-Protocol Directed Sedation Management on Mechanically Ventilated Patients in an Australian Intensive Care Unit.
Brief Title: Effectiveness of Sedation Management in an Australian Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: University of Melbourne (Other); Australian College of Critical Care Nurses (Other); Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2001.102
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Respiration Disorders
Keywords: sedation; mechanical ventilation; sedation protocols; critical care; intensive care outcomes; staffing
MeSH Terms: conditions — Respiration Disorders

INTERVENTIONS:
Procedure: Sedation management protocol

SUMMARY:
Sedation is an important treatment when caring for the critically ill patient on a respirator. Adequate sedation has been found to reduce stress, promote relaxation, induce amnesia, improve the tolerance of the respirator, and generally assist nursing care. However all sedation produces side effects for the patients. The aim of this study is to measure the effectiveness of two approaches to sedation management in an Australian Intensive Care unit.

DETAILED DESCRIPTION:
Sedation is an integral part of treatment in caring for the critically ill, ventilated patient. Adequate sedation has been found to reduce stress, promote relaxation, induce amnesia, improve the tolerance of ventilatory support, and generally assist nursing care. However, all the sedative agents produce significant side effects such as loss of consciousness, amnesia and haemodynamic instability. In view of the complex characteristics associated with sedative agents, it is important to systematically assess and evaluate their effectiveness in the clinical area. Two issues are important in determining the effective use of these agents. The first issue relates to the use of specific sedation scales to facilitate consistent interpretations among clinicians. The use of such scales is limited in Australia. The second issue relates to the practice of protocol-directed sedation. Despite support for decision-making tools to assist clinicians choice of sedative agents, few studies have evaluated their effectiveness. This research aims to compare the effectiveness of protocol-directed sedation management with traditional non protocol-directed practice in an Australian intensive care unit (ICU). In many Australian ICUs, the bedside nurse titrates the mechanical ventilation and sedation administration in consultation with the medical staff, usually in an unstructured manner.

This project builds upon a significant North American study that found a substantial decrease in the duration of mechanical ventilation, length of stay and rate of tracheostomy insertion following the implementation of a structured sedation protocol by nurses. However an exact replication of the protocol is not possible due to the lack of drug availability in Australia and the preferred drug regimes of RMH intensive care consultants. In addition, there are very few studies that document patients' memories of their experience being ventilated whilst sedated, despite documented discomfort such as anxiety, panic and difficulty synchronizing with the ventilator. There is a similar lack of literature on staff perceptions during the implementation of a multidisciplinary sedation protocol.

The research questions for this study are designed to examine three areas:

1. the differences between patients receiving protocol-directed sedation management compared with non protocol-directed sedation management;
2. the differences in patient perceptions of mechanical ventilation during protocol-directed sedation management as compared to non protocol-directed sedation management following extubation, and;
3. staff perceptions of using a sedation protocol in managing critically ill mechanically ventilated patients.

The design is a prospective, randomised, controlled trial studying 316 patients. There will be 158 patients recruited to the control group and 158 patients in the experimental group. The control group will receive the current management and the experimental group will receive protocol-directed sedation management. To explore patient perceptions of their experience, the patients will be interviewed using a semi-structured questionnaire following extubation and after receiving a rating of 4 on the sedation scale for 24 or more hours. In addition, staff perceptions will be surveyed on their attitudes and perceptions of the protocol.

This study will determine the efficacy and outcomes of protocol-directed sedation management of critically ill mechanically ventilated patients in an Australian context. The study will also improve our understanding of the patients' memories and perceptions during this period, which could lead to improved clinical practices and better patient outcomes. In understanding staff perceptions of the sedation protocol and its implementation, it will assist us to identify changes to improve education for new staff and compliance issues for ongoing implementation. It may be further useful in the future development of decision-making tools and their subsequent implementation and evaluation phases.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated

Exclusion Criteria:

* cardiac surgery patients
* those patients readmitted to the ICU who had been on the study during a previous admission were excluded for any subsequent admissions.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 316
Dates: Start 2001-11; Study Completion 2002-09

PRIMARY OUTCOMES:
Duration of Ventilation

SECONDARY OUTCOMES:
Length of stay
Tracheostomy insertion rate
Self extubation rate

CONTACTS AND LOCATIONS:
Overall Officials: Tracey K Bucknall, RN PhD, Principal Investigator — University of Melbourne
Locations (1):
- Royal Melbourne Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Result] Rose RL, Bucknall T. Staff perceptions on the use of a sedation protocol in the intensive care setting. Aust Crit Care. 2004 Nov;17(4):151-9. doi: 10.1016/s1036-7314(04)80020-1. PMID 18038524
- [Derived] Bucknall TK, Manias E, Presneill JJ. A randomized trial of protocol-directed sedation management for mechanical ventilation in an Australian intensive care unit. Crit Care Med. 2008 May;36(5):1444-50. doi: 10.1097/CCM.0b013e318168f82d. PMID 18434914